CLINICAL TRIAL: NCT03069326
Title: Evaluation of Ruxolitinib And Thalidomide Combination as a Therapy for Patients With Myelofibrosis
Brief Title: A Clinical Study to Test the Effects of Ruxolitinib And Thalidomide Combination for Patients With Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); Celgene (Industry); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1498
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Myelofibrosis
Keywords: Ruxolitinib; Thalidomide; 16-1498
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; Thalidomide

STUDY DESIGN:
Intervention Model Description: This is a multicenter, two stage phase II trial designed to assess the effect of ruxolitinib and thalidomide combination in subjects with Primary, Post Polycythemia Vera, or Post Essential Thrombocythemia Myelofibrosis (PMF, post-PV MF, or post-ET MF).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Ruxolitinib and Thalidomide (Experimental): After 3 cycles of ruxolitinib treatment, either prior to study enrollment or through the ruxolitinib run-in phase, patients who meet eligibility criteria will be treated with ruxolitinib and thalidomide orally on days 1-28 of a 28 day cycle. Cycles will be continued until the patient wishes to be removed from the study, unacceptable toxicity develops, disease progression, treating physician recommends removal, or termination of study occurs.
  Interventions: Drug: Ruxolitinib; Drug: Thalidomide
- Cohort B: Ruxolitinib and Thalidomide (Experimental): A cohort expansion, for patients with baseline thrombocytopenia, will enroll 35 additional patients
  After 3 cycles of ruxolitinib treatment, either prior to study enrollment or through the ruxolitinib run-in phase, patients who meet eligibility criteria will be treated with ruxolitinib and thalidomide orally on days 1-28 of a 28 day cycle. Cycles will be continued until the patient wishes to be removed from the study, unacceptable toxicity develops, disease progression, treating physician recommends removal, or termination of study occurs.
  Interventions: Drug: Ruxolitinib; Drug: Thalidomide

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib will be given orally in an outpatient setting unless the patient is being seen inpatient for another reason. Ruxolitinib will be given continuously orally daily in 28-day cycles.
Drug: Thalidomide — Thalidomide will be given orally in an outpatient setting unless the patient is being seen inpatient for another reason. thalidomide will be given continuously orally daily in 28-day cycles.

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drugs called ruxolitinib and thalidomide. Ruxolitinib and thalidomide could shrink the cancer, but it could also cause side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelofibrosis (either primary or post essential thrombocythemia/polycythemia vera) requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate-1 or -2 or high risk IPSS, DIPSS, DIPSS+, MIPSS70 or MIPSS70+ v2.0 score
* Patients taking Ruxolitinib at the time of enrollment must have been taking Ruxolitinib for a minimum of 3 months, and must have been on a stable dose of Ruxolitinib for a minimum of 4 weeks immediately prior to enrollment. However, for patients in the thrombocytopenic cohort A expansion, patients taking Ruxolitinib at the time of enrollment who are deemed to have a suboptimal response or are refractory to Ruxolitinib single-agent therapy (less than partial response per IWG criteria) must have been taking Ruxolitinib for a minimum of 6 weeks, and must have been on a stable dose of Ruxolitinib for a minimum of 4 weeks immediately prior to enrollment
* Patients taking Ruxolitinib at the time of enrollment must be deemed to have had a suboptimal response (less than partial response per IWG criteria) to Ruxolitinib single-agent therapy or deemed to have progression of disease (per IWG criteria).
* Age ≥ 18 years at the time of signing the informed consent.
* ECOG performance status 0 to 2.
* Patients must have adequate organ function as demonstrated by the following:

  1. Total bilirubin ≤ 2.0 mg/dL, unless due to Gilbert's disease
  2. Serum creatinine ≤ 2.0 mg/dL.
  3. ALT and AST ≤ 3 x upper limit of normal (unless the transaminitis is considered to be related to MF, in which case ≤5 x ULN is allowed
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 14 days prior to and again within 24 hours* of starting Thalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking Thalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* All study participants must be registered into the mandatory REMS® program, and be willing and able to comply with the requirements of REMS®
* Platelets ≥ 50000/uL and ANC ≥ 1000. For patients enrolled in the thrombocytopenic cohorts, platelet count must be >/= 25,000 but </= 99,000/uL.
* All study participants must be able to swallow oral medication

Exclusion Criteria:

* Use of any other standard anti-neoplastic drug or growth factor (e.g., anagrelide, G-CSF, revlimid, clofarabine) except hydroxyurea or experimental drugs, with the exception of Ruxolitinib, less than 14 days or 5-half lives prior to starting study therapy and/or lack of recovery from all toxicity from previous therapy to grade 1 or better.
* Known prior clinically relevant hypersensitivity reaction to Thalidomide, including the development of erythema nodosum if characterized by a desquamating rash.
* Prior therapy with Thalidomide in combination with Ruxolitinib
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form, which places the subject at unacceptable risk if he/she were to participate in the study or which confounds the ability to interpret data from the study.
* Pregnant or lactating females.
* Known positive for HIV or hepatitis B or C per institutional standard of care
* Participants with prior history of thromboembolic disease (i.e. deep venous thrombosis (DVT) or pulmonary embolism (PE) within the last six months, as Thalidomide has demonstrated an increased risk of DVT or PE
* Known to have a hypercoagulability syndrome (e.g.: antithrombin III, deficiency, anticardiolipin syndrome etc).
* Concurrent use of any strong inducers or strong inhibitors of CYP3A4. (See Appendix F for a list of prohibited and cautionary CYP3A4 inhibitors and inducers)
* Patients with active malignancy of other type than required for this study are not eligible with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
best objective response rate (ORR) | 1 year
  (ORR; complete response, partial response, and clinical improvement by IWG-MRT) in the first six cycles of the combination therapy. Clinical improvement for this endpoint will be defined as the change in anemia, spleen, and symptom response from the time of the initiation the combination therapy. The ORR will be defined as the best response by the completion of cycle 6 of combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Raajit Rampal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm